CLINICAL TRIAL: NCT03763500
Title: AMADEUS Atrial Fibrillation Monitoring in the Ablacure Database Including Patient-reported Outcomes and an Educational Program Used for Structured Care.
Brief Title: Evaluation of the Added Value of an Internet-based Educational Program for Patients With Atrial Fibrillation.
Acronym: AMADEUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulla Walfridsson (Other Government)
Collaborators: Dept of Internal Medicin, County Hospital Ryhov, Jönköping, Sweden. (Unknown); Dept of Cardiology, Örebro University Hospital, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Ulla Walfridsson, Principal investigator, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LiU Amadeus 2018
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation; Quality of Life; Signs and Symptoms; Health Economy
Keywords: Atrial fibrillation; Symptom burden; Health-related quality of life; Health economy
MeSH Terms: conditions — Atrial Fibrillation; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: prospective, randomized and open study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention): Regular care at participating hospitals:
  Extended written information and education of patients with atrial fibrillation.
- Internet-based education (Active Comparator): Patients randomized in this arm receive an Internet-based educational program in addition to extended written information. This includes 6 steps with detailed information on background, symptoms, investigations, treatment options, life-style as well as one part with guides to self management.
  Interventions: Other: Internet-based education

INTERVENTIONS:
Other: Internet-based education — A six-step Internet-based patient education.
  Arms: Internet-based education

SUMMARY:
This study is prospective, open and randomized concerning the value of an Internet-based educational program for patients with atrial fibrillation compared to "care as usual".

DETAILED DESCRIPTION:
In the present guidelines for treatment of atrial fibrillation education and information are underlined as important parts of the care. The investigators developed an Internet-based educational program in close collaboration with patients, specialists in the field, both physicians and nurses, and a phycologist, specialized in cognitive behavioral therapy.

The aim of the study is to evaluate this program in comparison to "care as usual" with reduction in symptom burden as primary endpoint, secondary endpoints being improvement in health-related quality of life and reduction in health-care costs.

ELIGIBILITY:
Inclusion Criteria:

Patients evaluated for electrical or pharmaceutical cardioversion or evaluated for treatment with antiarrhythmic drugs for paroxysmal or persistent atrial fibrillation.

Exclusion Criteria:

Age below 18, planned for cardiac surgery or catheter ablation, acute coronary syndrome during three months prior to randomisation. Insufficient knowledge of the Swedish language or other reasons making it impossible for the patient to independently fill out the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Symptom burden | One year after randomisation
  Arrhythmia related symptoms evaluated with the validated questionnaire ASTA (The Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmia)

SECONDARY OUTCOMES:
Health-related quality of life | One year after randomisation
  Arrhythmia related impact on health-related quality of life evaluated with the validated questionnaire ASTA (The Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmia)
Health economy | One year prior to and one year after randomisation
  Health-care costs during the year prior to the study and for the two arm during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Walfridsson, RN PhD, Study Chair — Dept of Cardiology, IMH, Linkoeping University, Sweden
Locations (3):
- Sweden (3):
  - Dept of Cardiology, University Hospital, Örebro, Närke
  - Dept of Internal Medicine, County Hospital, Jönköping, Småland
  - Dept of Cardiology, HMC, University Hospital, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No